CLINICAL TRIAL: NCT04512482
Title: A Visual Evaluation of Oral Plaque Removal Utilizing an Adjunct Enzyme Pre-rinse in Orthodontic Subjects
Brief Title: Evaluation of Oral Plaque Removal Utilizing an Adjunct Enzyme Pre-rinse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Water Pik, Inc. (Industry); Delta Dental Foundation (Other)
Responsible Party: Principal Investigator, Kelton Stewart, Chair & Program Director, Department of Orthodontics and, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1802369383
Record Dates: First submitted 2019-07-22; First posted 2020-08-13 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Dental Plaque; Dental Caries
Keywords: proteolytic enzyme; plaque removal; oral hygiene; orthodontic treatment
MeSH Terms: conditions — Dental Plaque; Dental Caries | interventions — Bromelains

STUDY DESIGN:
Intervention Model Description: Enrolled subjects undergoing orthodontic treatment with fixed appliances will be randomized to receive either the Bromelain rinse or Placebo first and then will be crossed over to receive the opposite intervention. The study will consist of two treatment period (1 day) separated by a washout period of 1 week.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Investigators were blinded during the clinical phase of the study and were unaware of the agents the subjects received. The investigators were also blinded during the visual plaque score analysis of the project and were unaware of what photograph corresponded to what phase or intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Bromelain, Then Placebo (Experimental): Subjects were asked to chew a disclosing tablet, swish, and expectorate. Intraoral photographs were obtained. They then received a vial containing 1 gram of bromelain that was reconstituted with 15ml of pineapple juice at 50 degrees F. Subjects swished the solution in their mouth for 2 minutes and then expectorated. Intraoral photographs were obtained. Subjects then received a toothbrush and were asked to brush their teeth for 2 minutes. Intraoral photographs were obtained. The subjects were then given a Waterpik and instructed to use the appliances to clean their teeth and brackets to the best of their ability, for 2 minutes. Intraoral photographs were obtained. After a 1 week washout period, they received the placebo rinse (powdered sugar), following the same protocol and series of intraoral photographs.
  Interventions: Drug: Bromelain; Other: Powdered sugar
- Experimental: Placebo, Then Bromelain (Placebo Comparator): Subjects were asked to chew a disclosing tablet, swish, and expectorate. Intraoral photographs were obtained. They then received a vial containing 1 gram of powdered sugar that was reconstituted with 15ml of pineapple juice at 50 degrees F. Subjects swished the solution in their mouth for 2 minutes and then expectorated. Intraoral photographs were obtained. Subjects then received a toothbrush and were asked to brush their teeth for 2 minutes. Intraoral photographs were obtained. The subjects were then given a Waterpik and instructed to use the appliances to clean their teeth and brackets to the best of their ability, for 2 minutes. Intraoral photographs were obtained. After a 1 week washout period, they received the bromelain rinse, following the same protocol and series of intraoral photographs.
  Interventions: Drug: Bromelain; Other: Powdered sugar

INTERVENTIONS:
Drug: Bromelain — The subjects were randomized to either receive the bromelain pre-rinse or the powdered sugar placebo pre-rinse. Subjects then had a 5-9 day washout period and was then exposed to the other intervention.
  Other Names: proteolytic enzyme rinse
Other: Powdered sugar — The subjects were randomized to either receive the bromelain pre-rinse or the powdered sugar placebo pre-rinse. Subjects then had a 5-9 day washout period and was then exposed to the other intervention.
  Other Names: placebo rinse

SUMMARY:
This study aims to investigate the impact of a bromelain pre-rinse adjunct on oral plaque removal in orthodontic subjects. The study's null hypothesis states that there is no statistically significant difference in visual plaque scores among orthodontic subjects with or without proteolytic enzyme rinse aid.

DETAILED DESCRIPTION:
Bromelain, a naturally occurring cysteine protease, from pineapple stalks, is used in food and medical industries and listed on the FDA's "Generally Recognized As Safe" (GRAS) list. In vitro bromelain study demonstrated antibacterial effect on oral pathogens. Bromelain was found to prevent biofilm formation by interfering with bacteria-bacteria adhesion and/or adhesion to enamel surface. Clinical trials with toothpaste containing bromelain demonstrated improved plaque and gingivitis scores and extrinsic enamel stain removal capabilities. The impact of bromelain application prior to traditional mechanisms of plaque removal have not been clearly evaluated.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* 10 to 25 years of age
* willing to consent to participation
* able to follow study instructions
* in active orthodontic treatment with fixed orthodontic appliances

Exclusion Criteria:

* unwilling/unable to follow study instructions
* documented/suspected pineapple allergy
* proteolytic enzyme allergy
* food dye allergy
* smoker

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelton Stewart, DDS, MS, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred from 6/14/2018 to 7/3/2018 from the graduate orthodontic clinic in the Indiana University School of Dentistry. 46 patients were screened for eligibility during this time frame.
Pre-assignment Details: 46 of 46 subjects were randomized. Of those, 45 subjects completed at least one of the two study interventions (one of the study arms).
Groups:
- Placebo & Bromelain: Subjects were asked to chew a disclosing tablet, swish, and expectorate. Intraoral photographs were obtained. They then received a vial containing 1 gram of powdered sugar that was reconstituted with 15ml of pineapple juice at 50 degrees F. Subjects swished the solution in their mouth for 2 minutes and then expectorated. Intraoral photographs were obtained. Subjects then received a toothbrush and were asked to brush their teeth for 2 minutes. Intraoral photographs were obtained. The subjects were then given a Waterpik and instructed to use the appliances to clean their teeth and brackets to the best of their ability, for 2 minutes. Intraoral photographs were obtained.
  Subjects completed a 1 week (5-9 day) washout period and then completed the protocol again but received the bromelain rinse.
- Bromelain & Placebo: Subjects were asked to chew a disclosing tablet, swish, and expectorate. Intraoral photographs were obtained. They then received a vial containing 1 gram of bromelain that was reconstituted with 15ml of pineapple juice at 50 degrees F. Subjects swished the solution in their mouth for 2 minutes and then expectorated. Intraoral photographs were obtained. Subjects then received a toothbrush and were asked to brush their teeth for 2 minutes. Intraoral photographs were obtained. The subjects were then given a Waterpik and instructed to use the appliances to clean their teeth and brackets to the best of their ability, for 2 minutes. Intraoral photographs were obtained.
  Subjects completed a 1 week (5-9 day) washout period and then completed the protocol again but received the placebo (powdered sugar).
Period: First Intervention (1 Day)
Arm/Group | Placebo & Bromelain | Bromelain & Placebo
Started | 24 | 21
Baseline Plaque Assessment | 24 | 21
Baseline Photographs | 24 | 21
Received Rinse Intervention | 24 | 21
Post-rinse Photographs | 24 | 21
Toothbrush Utilization | 24 | 21
Post-toothbrush Photographs | 24 | 21
Waterpik Utilization | 24 | 21
Post-Waterpik Photographs | 24 | 21
Completed | 24 | 21
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Placebo & Bromelain | Bromelain & Placebo
Started | 24 | 21
Completed | 24 | 21
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Placebo & Bromelain | Bromelain & Placebo
Started | 24 | 21
Baseline Plaque Assessment | 22 | 20
Baseline Photographs | 22 | 20
Received Intervention | 22 | 20
Post-rinse Photographs | 22 | 20
Toothbrush Utilization | 22 | 20
Post-toothbrush Photographs | 22 | 20
Waterpik Utilization | 22 | 20
Post-Waterpik Photographs | 22 | 20
Completed | 22 | 20
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo & Bromelain: Subjects were asked to chew a disclosing tablet, swish, and expectorate. Intraoral photographs were obtained. They then received a vial containing 1 gram of powdered sugar (placebo) that was reconstituted with 15ml of pineapple juice at 50 degrees F. Subjects swished the solution in their mouth for 2 minutes and then expectorated. Intraoral photographs were obtained. Subjects then received a toothbrush and were asked to brush their teeth for 2 minutes. Intraoral photographs were obtained. The subjects were then given a Waterpik and instructed to use the appliances to clean their teeth and brackets to the best of their ability, for 2 minutes. Intraoral photographs were obtained.
  Subjects then had a 1 week (5-9 day) washout period and were then exposed to the other intervention (bromelain rinse).
- Bromelain & Placebo: Subjects were asked to chew a disclosing tablet, swish, and expectorate. Intraoral photographs were obtained. They then received a vial containing 1 gram of bromelain that was reconstituted with 15ml of pineapple juice at 50 degrees F. Subjects swished the solution in their mouth for 2 minutes and then expectorated. Intraoral photographs were obtained. Subjects then received a toothbrush and were asked to brush their teeth for 2 minutes. Intraoral photographs were obtained. The subjects were then given a Waterpik and instructed to use the appliances to clean their teeth and brackets to the best of their ability, for 2 minutes. Intraoral photographs were obtained.
  Subjects then had a 1 week (5-9 day) washout period and were then exposed to the other intervention (placebo rinse).
- Total: Total of all reporting groups
Arm/Group | Placebo & Bromelain | Bromelain & Placebo | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 16 | 35
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 11 | 9 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Composite Plaque Score
Description: The composite plaque score refers to the cumulative plaque score of all twelve teeth following the administration of the bromelain and placebo (powdered sugar) solutions. The composite plaque score scale had a minimum value of 0 and a maximum value of 48. A score of 0 indicated no plaque was observed on the teeth, while a a score of 48 indicated severe plaque on all possible tooth surfaces. A lower plaque score reflects a better outcome, while a higher plaque score a worse outcome.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bromelain: Subjects were asked to chew a disclosing tablet, swish, and expectorate. Intraoral photographs were obtained. They then received a vial containing 1 gram of bromelain that was reconstituted with 15ml of pineapple juice at 50 degrees F. Subjects swished the solution in their mouth for 2 minutes and then expectorated. Intraoral photographs were obtained. Subjects then received a toothbrush and were asked to brush their teeth for 2 minutes. Intraoral photographs were obtained. The subjects were then given a Waterpik and instructed to use the appliances to clean their teeth and brackets to the best of their ability, for 2 minutes. Intraoral photographs were obtained.
  Bromelain: The subjects were randomized to either receive the bromelain pre-rinse or the powdered sugar placebo pre-rinse. Subjects then had a 5-9 day washout period and was then exposed to the other intervention.
- Placebo: Subjects were asked to chew a disclosing tablet, swish, and expectorate. Intraoral photographs were obtained. They then received a vial containing 1 gram of powdered sugar that was reconstituted with 15ml of pineapple juice at 50 degrees F. Subjects swished the solution in their mouth for 2 minutes and then expectorated. Intraoral photographs were obtained. Subjects then received a toothbrush and were asked to brush their teeth for 2 minutes. Intraoral photographs were obtained. The subjects were then given a Waterpik and instructed to use the appliances to clean their teeth and brackets to the best of their ability, for 2 minutes. Intraoral photographs were obtained.
  Powdered sugar: The subjects were randomized to either receive the bromelain pre-rinse or the powdered sugar placebo pre-rinse. Subjects then had a 5-9 day washout period and was then exposed to the other intervention.
Arm/Group | Bromelain | Placebo
Number analyzed (Participants) | 43 | 43
score on a scale | 36.2 (10.7) | 37.9 (10.8)
Statistical Analysis 1: Comparison: Bromelain vs Placebo; A power analysis determined that a sample size of forty-five (45) subjects would possess 90% power to detect an effect size of 0.5 between the intervention and control legs of the crossover design. With 43 total subjects the study had between 85 and 90% power; Test type: Superiority; p = .044, ANOVA

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Bromelain | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT04512482/Prot_SAP_001.pdf